CLINICAL TRIAL: NCT00303316
Title: Immunogenicity Study of the Antibody Persistence and Booster Effect of PENTAXIM™ at 18 Months of Age Following a Primary Series of DTaP-IPV-HB-PRP~T Combined Vaccine or of PENTAXIM™ and ENGERIX B® PEDIATRICO at 2, 4, and 6 Months of Age in Healthy Argentinean Infants
Brief Title: Immunogenicity Study of Antibody Persistence and Booster Effect of PENTAXIM™ at 18 Months in Healthy Argentinean Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A3L16
Record Dates: First submitted 2006-03-13; First posted 2006-03-16 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-01

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis; Hepatitis B
Keywords: Diphtheria; Tetanus; Pertussis; whooping cough; Haemophilus influenzae type b; Hepatitis B; Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Hepatitis B; Haemophilus Infections | interventions — Pentavac

ARMS (2):
- DTacP IPV HepB PRP-T Combined Vaccine Group (Experimental): Participant will receive a booster dose of PENTAXIM™ having received DTacP-IPV-HepB-PRP-T (primary series) in Study A3L02.
  Interventions: Biological: DTaP-IPV//PRP~T combined vaccine
- PENTAXIM™ and ENGERIX B® Vaccine Group (Active Comparator): Participant will receive a booster dose of PENTAXIM™ having received ENGERIX B® and PEDIATRICO in Study A3L02 (Primary series)
  Interventions: Biological: DTaP-IPV//PRP~T combined vaccine

INTERVENTIONS:
Biological: DTaP-IPV//PRP~T combined vaccine — 0.5 mL, Intramuscular
  Other Names: PENTAXIM™
  Arms: DTacP IPV HepB PRP-T Combined Vaccine Group
Biological: DTaP-IPV//PRP~T combined vaccine — 0.5 mL, Intramuscular
  Other Names: PENTAXIM™
  Arms: PENTAXIM™ and ENGERIX B® Vaccine Group

SUMMARY:
This study will assess both the antibody persistence of the investigational vaccine and the immune response and safety of a booster dose of PENTAXIM™ vaccine in 18 months-old toddlers who participated in an earlier study in order to determine if they are still protected before they receive a booster dose of D, T, IPV, pertussis or Hib vaccines and also to assess the quality of the induced immune memory in response to a booster dose of the same vaccine as in the primary series.

Primary Objective:

To describe the antibody persistence at 18 months of age and the booster effect of a dose of PENTAXIM™ on immunogenicity.

Secondary objective:

To describe the safety profile of the booster dose PENTAXIM™ in each vaccine group defined by the vaccines received during the primary series.

ELIGIBILITY:
Inclusion Criteria:

* Toddler at 18 months of age (range: 510 days to 578 days of age inclusive)
* Participated in study A3L02 (NCT00831311) and has completed the three-dose primary series with either diphtheria, tetanus, pertussis (2-component acellular), recombinant Hepatitis B Hansenula and poliomyelitis vaccine adsorbed, and Haemophilus influenzae type b vaccine, conjugated to tetanus protein (DTaP-IPV-HB-PRP~T) or PENTAXIM™ and ENGERIX B® PEDIATRICO at 2, 4, and 6 months of age
* Written informed consent form signed by at least one parent or by a legal representative and an independent witness
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial in the four weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months or long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the last six months
* Any vaccination in the four weeks preceding the trial
* Vaccination with a vaccine containing diphtheria, tetanus, pertussis, Haemophilus influenzae type b, polio, or hepatitis B antigen, since the end of the primary series
* History of documented diphtheria, tetanus, pertussis, Haemophilus influenzae type b, polio, or hepatitis B infection(s) (confirmed either clinically, serologically, or microbiologically)
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* History of seizures
* Fever (axillary temperature ≥37.4°C or equivalent rectal temperature ≥38.0°C) or acute illness on the day of inclusion
* Known contraindication to further vaccination with a pertussis vaccine such as:
* Encephalopathy; Inconsolable crying for >3 hours within 48 hours following vaccine injection
* Hypotonic hyporesponsive episode within 48 hours following vaccine injection
* Seizures with or without fever within three days following vaccine injection
* Axillary temperature >39.4°C or equivalent rectal temperature > 40.0°C within 48 hours following vaccine injection.

Ages: 510 Days to 578 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 458 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Córdoba, Córdoba Province, Argentina

REFERENCES:
- [Result] Tregnaghi M, Zambrano B, Santos-Lima E. Antibody persistence after a primary series of a new DTaP-IPV-Hep B-PRP-T combined vaccine or separate DTaP-IPV//PRP-T and hepatitis B vaccines at 2, 4, and 6 months of age and the effect of a subsequent DTaP-IPV//PRP-T booster vaccination at 18 months of age in healthy Argentinean infants. Pediatr Infect Dis J. 2012 Jan;31(1):e24-30. doi: 10.1097/INF.0b013e318242460a. PMID 22157567
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 February 2006 to 03 October 2006 at 1 clinical center in Argentina.
Pre-assignment Details: A total of 458 participants who met all the inclusion and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- DTacP-IPV-Hep B-PRP~T Group: Participants received a booster dose of PENTAXIM™ at 18 months of age in this study. They had received 3 primary-series doses of Diphtheria (D), Tetanus (T), Pertussis (acellular component [aP]), hepatitis B (Hep B [recombinant DNA]) and poliomyelitis (Inactivated [IPV]), and Haemophilus influenzae type b (Hib) conjugated vaccine adsorbed (DTaP-IPV-HepB-PRP~T), (1 dose each at 2, 4, and 6 months of age) in Study A3L02 (NCT00831311).
- PENTAXIM™ and ENGERIX B® Group: Participants received a booster dose of PENTAXIM™ at 18 months of age in this study. They had received 3 primary-series doses of PENTAXIM™ and ENGERIX B® PEDIATRICO (1 dose each at 2, 4, and 6 months of age) in Study A3L02 (NCT00831311).
Period: Overall Study
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group
Started | 232 | 226
Completed | 230 | 223
Not Completed | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group | Total
Number analyzed (Participants) | 232 | 226 | 458
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 232 | 226 | 458
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Months] | 17.6 (0.436) | 17.7 (0.492) | 17.6 (0.465)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 214
  Male | 125 | 119 | 244
Region of Enrollment [Number; unit: Participants]
  Argentina | 232 | 226 | 458

OUTCOME MEASURES:

1. Primary Outcome: Summary of Antibody Persistence at 18 Months of Age in Participants That Received Primary Series Vaccination of Either DTaP-IPV-HepB-PRP~T or PENTAXIM™ and ENGERIX B® PEDIATRICO at 2, 4, and 6 Months of Age.
Description: Antibody persistence (pre-booster) were defined as titers ≥ 10 mIU/mL for hepatitis B (Hep B;); ≥ 0.15 µg/mL for Haemophilus influenzae type b (PRP); ≥ 0.01 IU/mL for Diphtheria and Tetanus; ≥ 8 (1/dil) for polio types 1, 2, and 3; and ≥ 4 EU/mL for Pertussis Toxoid (PT) and Filamentous Hemagglutinin (FHA).
Time Frame: Day 0 (Before booster vaccination)
Population: Antibody Persistence was assessed in all enrolled participants with pre-booster vaccination data (Intent-to-Treat population).
Measure: Number; unit: Participants
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group
Number analyzed (Participants) | 232 | 226
Participants
  Anti-Hepatitis B (N = 228, 222) | 195 | 221
  Anti-PRP (N = 224, 217) | 171 | 164
  Anti-Diphtheria (N = 228, 221) | 169 | 165
  Anti-Tetanus (N = 229, 216) | 229 | 216
  Anti-Polio 1 (N = 214, 205) | 213 | 205
  Anti-Polio 2 (N = 217, 204) | 215 | 203
  Anti-Polio 3 (N = 214, 203) | 205 | 199
  Anti-Pertussis Toxoid (N= 216, 212) | 190 | 190
  Anti-Filamentous Hemagglutinin (N = 230, 220) | 228 | 213

2. Primary Outcome: Summary of Booster Response in Participants at 18 Months of Age Following Booster Vaccination With PENTAXIM™ Following a Primary Series Vaccination of Either DTaP-IPV-HepB-PRP~T or PENTAXIM™ and ENGERIX B® PEDIATRICO at 2, 4, and 6 Months of Age.
Description: Booster response were defined as titers ≥ 1.0 µg/mL for Haemophilus influenzae type b (PRP); ≥ 0.1 IU/mL for Diphtheria and Tetanus; ≥ 8 (1/dil) for Polio types 1, 2, and 3; and for Pertussis Toxoid (PT) and Filamentous Hemagglutinin (FHA) ≥ 4 EU/mL and a ≥ 4 fold increase from pre-booster to post-booster value.
Time Frame: Day 30 Post-booster Vaccination
Population: Booster responses were assessed in all vaccinated participants with endpoint data following the booster vaccination (Intent-to-Treat population).
Measure: Number; unit: Participants
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group
Number analyzed (Participants) | 232 | 226
Participants
  Anti-PRP (N = 223, 216) | 220 | 215
  Anti-Diphtheria (N = 225, 221) | 216 | 214
  Anti-Tetanus (N = 222, 219) | 222 | 219
  Anti-Polio 1 (N = 211, 209) | 211 | 209
  Anti-Polio 2 (N = 208, 210) | 208 | 210
  Anti-Polio 3 (N = 205, 205) | 205 | 205
  Anti-Pertussis Toxoid (N = 226, 220) | 226 | 220
  Anti-Pertussis Toxoid (4-Fold Rise: N = 211, 208) | 202 | 199
  Anti-Filamentous Hemagglutinin (N = 227, 221) | 227 | 221
  Anti-FHA (4-Fold Rise: N = 225, 215) | 198 | 202

3. Secondary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Post-booster Vaccination With PENTAXIM™
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, Irritability.
  Grade 3 was defined as: Pain, cries when injected limb is moved or movement of limb is reduced; Erythema and Swelling, ≥ 5 cm; Pyrexia, ≥ 39.6ºC; Vomiting, ≥ 6 episodes/24 hour or requiring parenteral hydration; Crying, > 3 hours; Somnolence, sleeping most of the time or difficulty to wake up; Anorexia, refuses ≥ 3 feeds/meals or refuses most feeds/meals; and Irritability, inconsolable.
Time Frame: Day 0 up to Day 30 post-booster vaccination
Population: Solicited injection site and systemic reactions were assessed in the enrolled and vaccinated participants, Safety Analysis Set population.
Measure: Number; unit: Participants
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group
Number analyzed (Participants) | 231 | 223
Participants
  Injection site Pain | 112 | 117
  Grade 3 Injection site Pain | 8 | 12
  Injection site Erythema | 66 | 93
  Grade 3 Injection site Erythema | 7 | 19
  Injection site Swelling | 63 | 89
  Grade 3 Injection site Swelling | 5 | 20
  Any Pyrexia | 47 | 44
  Grade 3 Pyrexia | 9 | 4
  Any Vomiting | 18 | 18
  Grade 3 Vomiting | 0 | 0
  Any Crying | 61 | 53
  Grade 3 Crying | 3 | 2
  Any Somnolence | 52 | 44
  Grade 3 Somnolence | 6 | 2
  Any Anorexia | 59 | 52
  Grade 3 Anorexia | 9 | 3
  Any Irritability | 85 | 78
  Grade 3 Irritability | 6 | 1

4. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Before and After Booster Vaccination With PENTAXIM™ Following a Primary Series Vaccination of Either DTaP-IPV-HepB-PRP~T or PENTAXIM™ and ENGERIX B® PEDIATRICO at 2, 4, and 6 Months of Age.
Description: Antibody titers determination:
  Hepatitis B (Hep B) by enhanced chemiluminescence assay; Haemophilus influenzae type b (PRP), Tetanus, Pertussis toxoid (PT) and filamentous hemagglutinin (FHA) by enzyme linked immunosorbent assay (ELISA); Diphtheria by neutralization test; Poliovirus types 1,2, and 3 by microneutralization assay.
Time Frame: Day 0 (pre-booster) and Day 30 post-booster
Population: Geometric mean titers were assessed in all participants with endpoint data who received the booster vaccine (Intent-to-Treat Analysis Set for immunogenicity).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group
Number analyzed (Participants) | 232 | 226
Titers
  Anti-Hepatitis B Pre-booster (N = 228, 222) | 87.6 [69.2 to 111] | 197 [168 to 230]
  Anti-PRP Pre-booster (N = 224, 217) | 0.399 [0.327 to 0.487] | 0.326 [0.270 to 0.394]
  Anti-PRP Post-booster (N = 223, 216) | 27.4 [23.0 to 32.7] | 41.4 [35.0 to 48.8]
  Anti-Diphtheria Pre-booster (N = 228, 221) | 0.022 [0.018 to 0.027] | 0.018 [0.015 to 0.022]
  Anti-Diphtheria Post-booster (N = 225, 221) | 1.92 [1.58 to 2.32] | 2.11 [1.74 to 2.56]
  Anti-Tetanus Pre-booster (N = 229, 216) | 0.287 [0.255 to 0.325] | 0.171 [0.153 to 0.192]
  Anti-Tetanus Post-booster (N = 222, 219) | 4.81 [4.37 to 5.31] | 4.54 [4.07 to 5.08]
  Anti-Polio 1 Pre-booster (N= 214, 205) | 303 [251 to 365] | 232 [193 to 279]
  Anti-Polio 1 Post-booster (N = 211, 209) | 7243 [6218 to 8436] | 9996 [8521 to 11725]
  Anti-Polio 2 Pre-booster (N = 217, 204) | 370 [300 to 457] | 292 [234 to 366]
  Anti-Polio 2 Post-booster (N = 208, 210) | 8512 [7281 to 9952] | 11229 [9574 to 13170]
  Anti-Polio 3 Pre-booster (N = 214, 203) | 257 [202 to 327] | 223 [174 to 284]
  Anti-Polio 3 Post-booster (N = 205, 205) | 10975 [9066 to 13286] | 14482 [12067 to 17380]
  Anti-PT Pre-booster (N = 216, 212) | 10.7 [9.37 to 12.3] | 12.9 [11.3 to 14.7]
  Anti-PT Post-booster (N = 226, 220) | 226 [205 to 249] | 325 [292 to 362]
  Anti-FHA Pre-booster (N = 230, 220) | 28.2 [24.5 to 32.5] | 19.0 [16.7 to 21.6]
  Anti-FHA Post-booster (N = 227, 221) | 335 [305 to 368] | 333 [305 to 363]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (before booster vaccination) up to Day 30 post-booster vaccination in the Safety Analysis Set population.
Description: The Safety Analysis Set (SafAS) was defined as the set of participants who received the booster vaccine. The analysis was based upon the number of participants for whom each safety assessment was performed.
Arm/Group | DTacP-IPV-Hep B-PRP~T Group | PENTAXIM™ and ENGERIX B® Group
Serious Adverse Events (participants affected / at risk) | 3/231 | 1/223
Other Adverse Events (participants affected / at risk) | 134/231 | 137/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTacP-IPV-Hep B-PRP~T Group (N=231) | PENTAXIM™ and ENGERIX B® Group (N=223)
Otitis Media Acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTacP-IPV-Hep B-PRP~T Group (N=231) | PENTAXIM™ and ENGERIX B® Group (N=223)
Vomiting (Gastrointestinal disorders) | 18 (18) | 18 (18)
Solicited Injection Site Erythema (General disorders) | 66 (66) | 93 (93)
Solicited Injection Site Pain (General disorders) | 112 (112) | 117 (117)
Solicited Injection Site Swelling (General disorders) | 63 (63) | 89 (89)
Irritability (General disorders) | 85 (85) | 78 (78)
Pyrexia (General disorders) | 47 (47) | 44 (44)
Bronchitis (Infections and infestations) | 16 (16) | 8 (8)
Rhinitis (Infections and infestations) | 15 (15) | 14 (14)
Anorexia (Metabolism and nutrition disorders) | 59 (59) | 52 (52)
Somnolence (Nervous system disorders) | 52 (52) | 44 (44)
Crying (Psychiatric disorders) | 61 (61) | 53 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.